CLINICAL TRIAL: NCT06464328
Title: The Impact of Tai Chi Combined With Music Therapy Intervention on Depression and Anxiety Among College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiarun (Other)
Responsible Party: Sponsor-Investigator, Wu Jiarun, Principal Investigator, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: USM/JEPeM/22040247
Record Dates: First submitted 2024-06-02; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Unrecognized Condition
Keywords: Tai Chi combined with music therapy; depression; anxiety; college students
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi Combined with Music Therapy Intervention (Experimental): Tai Chi combined with music therapy Intervention, the effect was achieved by replacing the school's physical education classes with Tai Chi of the researchers' choice, and then by playing music of the researchers' choice during class.
  Interventions: Behavioral: Tai Chi Combined with Music Therapy Intervention
- Music intervention only (Experimental): Music only (the fast tempo of 120-130 bpm music will be selected) The effect was achieved by playing music selected by the researchers during originally physical education classes in school.
  Interventions: Behavioral: Music intervention only
- Tai Chi intervention only (Experimental): Tai Chi intervention only The effect was achieved by replacing the school's originally physical education classes with Tai Chi of the researchers' choice.
  Interventions: Behavioral: Tai Chi intervention only

INTERVENTIONS:
Behavioral: Tai Chi Combined with Music Therapy Intervention — Tai Chi combined with music therapy Intervention, the effect was achieved by replacing the school's physical education classes with Tai Chi of the researchers' choice, and then by playing music of the researchers' choice during class; twice a week for twelve weeks
  Arms: Tai Chi Combined with Music Therapy Intervention
Behavioral: Music intervention only — Music only (120-130 bpm) The effect was achieved by playing music selected by the researchers during originally physical education classes in school; twice a week for twelve weeks
  Arms: Music intervention only
Behavioral: Tai Chi intervention only — Tai Chi intervention only The effect was achieved by replacing the school's originally physical education classes with Tai Chi of the researchers' choice; twice a week for twelve weeks
  Arms: Tai Chi intervention only

SUMMARY:
This study aims to investigate the effects of Tai Chi combined with music therapy on alleviating depression and anxiety among college students. Depression and anxiety are prevalent among college students and have a significant impact on their lives and academic performance. Therefore, exploring effective interventions is crucial for promoting the mental health of college students.

ELIGIBILITY:
Inclusion Criteria:

* This study were being enrolled as a student at Tianjin University of Sport
* aged between 18 and 25 years
* proficient in reading and communicating in Chinese.

Exclusion Criteria:

* Students with visual impairments
* Students with auditory
* Students with other impairments

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Change from the Self-Rating Depression Scale (SDS) at week 12 | 12 weeks
  The SDS, developed by American researchers Zung (1965), is specifically designed to evaluate the degree of depression in participants. The survey comprises 20 items, and participants express their feelings using a Likert scale ranging from 1 (Never) to 4 (Always). The SDS has been widely utilized worldwide to measure depression levels, demonstrating strong internal consistency and validity (Cronbach's Alpha = 0.832), and has been well-established in clinical and research settings (Campo-Arias et al., 2006).
Change from the Self-Rating Anxiety Scale (SAS) at week 12 | 12 weeks
  The SAS developed by American researchers Zung, (2013), is tailored to assess the anxiety level of participants. This instrument consists of a concise 20-item questionnaire, and participants use a Likert scale ranging from 1 (Strongly Disagree) to 4 (Strongly Agree) to express their emotions. The SAS exhibits robust psychometric properties in assessing participants' anxiety levels, with acceptable reliability values. The internal consistency, measured through Cronbach's Alpha, is 0.897, and the test-retest reliability, represented by the intra-class correlation coefficient (ICC), is 0.913 (Samakouri et al., 2012).

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia